CLINICAL TRIAL: NCT03445806
Title: IOP Monitoring After Trabeculectomy Using iCare Home
Status: Terminated | Type: Observational
Why Stopped: Difficulty recruiting patients
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Enping Chen, Principal Investigator, St. Erik Eye Hospital
Other Study IDs: Home Trab
Record Dates: First submitted 2018-02-15; First posted 2018-02-26 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma, Open-Angle; Pseudo Exfoliation Syndrome
Keywords: IOP fluctuations; iCare Home; Trabeculectomy; self-tonometry
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate how much trabeculectomy influences intraocular pressure (IOP) fluctuations measured with iCare Home rebound tonometry (RTHome) in patients with primary open-angle glaucoma (POAG) or pseudo-exfoliation glaucoma (PEX).

DETAILED DESCRIPTION:
Fifty glaucoma patients (POAG and PEX) planned for trabeculectomy will be recruited.

At baseline, patients will be trained to use the iCare Home tonometer (RTHome), a handheld device based on rebound tonometry and designed for patients to use at home. After the training session and when patients feel confident, a measurement will be recorded. At the same visit, a new measurement will be obtained by the study staff, an optometrist or a nurse, using the same device. No IOP values will be visible for the examiner at that point. A single IOP measurement will be obtained by the same study staff using Goldmann applanation tonometry (GAT). Patients will come for a second visit where new measurements will be made in the same way as at baseline.

In between visits, patients will borrow the iCare Home tonometer to measure their IOP at 06 and 10 am, and at 2, 6 and 10 pm during three consecutive days to obtain an IOP curve.

Two-three months after trabeculectomy, a new IOP curve will be obtained following the same procedure as pre-operatively. There will be no restrictions in patients' daily activities regarding diet, physical activity or slee. If patients use any eyedrops, they will continue to use them as prescribed.

ELIGIBILITY:
Inclusion Criteria:

* POAG
* PXG

Exclusion Criteria:

* previous trabeculectomy
* reduced hand and arm mobility (e. due to rheumatism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive male and female patients, older than 18 y.o., at St Erik's Eye Hospital in Stockholm, Sweden, diagnosed with POAG or PXG and listed for a trabeculectomy.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Lowering of IOP levels after trabeculectomy | 2-3 months
  Mean (SD) IOP pre- and post trabeculectomy

SECONDARY OUTCOMES:
Lowering of IOP fluctuations after trabeculectomy | 2-3 months
  Mean (SD) IOP range pre- and post trabeculectomy

CONTACTS AND LOCATIONS:
Locations (1):
- St Erik Eye Hospital, Stockholm, Sweden